CLINICAL TRIAL: NCT01679119
Title: A Randomised Phase II Trial of Inotuzumab Ozogamicin Plus Rituximab & CVP (IO-R-CVP) vs Gemcitabine Plus Rituximab & CVP (Gem-R-CVP) for the First Line Treatment of Patients With DLBCL Who Are Not Suitable for Anthracycline Containing Chemotherapy
Brief Title: Treatment of Patients With Diffuse Large B Cell Lymphoma Who Are Not Suitable for Anthracycline Containing Chemotherapy
Acronym: INCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Pfizer (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL 11/0475
Record Dates: First submitted 2012-07-23; First posted 2012-09-05 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse large b cell lymphoma; Inotuzumab Ozogamicin; Gemcitabine; Rituximab; Cyclophosphamide; Vincristine; Prednisolone
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Vincristine; Prednisolone; Rituximab; Inotuzumab Ozogamicin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IO-R-CVP (Experimental): Inotuzumab Ozogamicin plus Rituximab and CVP (Cyclophosphamide, vincristine & prednisolone).
  Interventions: Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisolone; Drug: Rituximab; Drug: Inotuzumab Ozogamicin
- Gem-R-CVP (Active Comparator): Gemcitabine plus Rituximab and CVP (Cyclophosphamide, Vincristine and Prednisolone).
  Interventions: Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisolone; Drug: Rituximab; Drug: Gemcitabine

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 750mg/m2 IV, given day 1
Drug: Vincristine — Vincristine 1.4mg/m2(max 2mg)IV given day 1
Drug: Prednisolone — Prednisolone 100mg OD Oral given days 1-5
Drug: Rituximab — Rituximab 375mg/m2 IV given day 1
  Other Names: MabThera
Drug: Inotuzumab Ozogamicin — Inotuzumab Ozogamicin 0.8mg/m2 IV given on day 2
  Arms: IO-R-CVP
Drug: Gemcitabine — Gemcitabine up to 1g/m2 IV given day 1 and day 8 (Patients with ECOG PS 0-1: starting dose: 875mg/m2 (1st cycle). If tolerated can be escalated to 1g/m2 in cycle 2 and subsequent cycles. Patients with ECOG PS 2: starting dose 750mg/m2 (1st cycle). If tolerated can be escalated to 875mg/m2 in cycle 2 and then escalated to 1g/m2 in cycle 3 and subsequent cycles.)
  Arms: Gem-R-CVP

SUMMARY:
The purpose of this trial is to compare the efficacy and safety of Inotuzumab Ozogamicin in combination with R-CVP with that of R-G-CVP for the treatment of Diffuse Large B Cell Lymphoma (DLBCL) in a population of patients not suitable for anthracycline based chemotherapy.

There is no standard of care for the treatment of this group of patients. If demonstrated to be efficacious and safe to deliver this regimen will be further tested in a phase III trial to determine whether this should become the standard of care amongst patients with DLBCL not fit for anthracycline (R-CHOP).

DETAILED DESCRIPTION:
The incidence of DLBCL is increasing and with an expanding elderly population, the incidence will continue to rise. Given that about 40% of cases of DLBCL occur in patients aged over 70 and the number of co-mobilities increases with age, research to investigate the optimal treatment of DLBCL in this group of patients is needed. R-CHOP remains the standard of care for the majority of patients with DLBCL, anthracycline use is precluded in a proportion of these patients by a high risk of developing cardiotoxicity, especially congestive cardiac failure. Currently there is no standard of care for patients who are unfit for anthracycline treatment. It has been routine to omit the doxorubicin from R-CHOP, giving R-CVP instead. However the outcome for patients treated with R-CVP is poor and attempts have been made to replace the doxorubicin with alternative agents. The trial will compare an experimental arm consisting of Inotuzumab Ozogamicin added to the standard immunochemotherapy regimen of rituximab, cyclophosphamide, vincristine and prednisolone (R-CVP) with the control arm of gemcitabine added to the same combination (Gem-R-CVP).

ELIGIBILITY:
Inclusion criteria:

* Informed written consent for the trial
* Histologically proven diffuse large B cell lymphoma (DLBCL) according to the current World Health Organisation (WHO) classification including all morphological variants. The B cell nature of the proliferation must be verified by demonstration of CD20 positivity. A concurrent (synchronous) diagnosis of low grade lymphoma (e.g. on bone marrow trephine or presence of both low grade and DLBCL in a lymph node biopsy) or previous diagnosis of low grade lymphoma which hasn't been treated with a systemic therapy is permitted
* Bulky Stage IA (lymph node or lymph node mass ≥ 10cm in maximum diameter), stage IB, stage II, stage III and stage IV disease
* ECOG performance status 0-2
* Measurable disease
* Age 18 ≥ years
* Adequate contraceptive precautions for all patients of childbearing potential
* History of malignant disease diagnosed at any time in the past with completed radical treatment and the risk of relapsing within the next 5 years is <10%. Patients previously treated should be free of sequelae of treatment which would compromise the delivery of study drugs as compared with other eligible patients.
* No previous chemotherapy, radiotherapy or other investigational drug for this indication - previous corticosteroids up to a dose equivalent to prednisolone 1mg/kg/day for up to 14 days are permitted prior to randomisation EITHER
* Unsuitable for anthracycline-containing chemotherapy due to impaired cardiac function defined by an ejection fraction of ≤ 50% OR Left ventricle ejection fraction > 50% but in the presence of significant co-morbidities (diabetes mellitus, hypertension or ischaemic heart disease) precluding anthracycline-containing chemotherapy as determined by treating physician. Co-morbidities must be documented on the randomisation form and CIRS score recorded
* Adequate bone marrow function (Platelets > 100x109/l, WBC > 3.0x109/l, Neutrophils > 1.5x109/l) at time of study entry unless attributed to bone marrow infiltration by DLBCL
* Life expectancy > 3 months

Exclusion criteria:

* Symptomatic central nervous system or meningeal involvement by DLBCL
* Previous diagnosis of low grade lymphoma which has been treated with a systemic therapy
* Non-bulky stage IA disease
* ECOG performance status 3-4
* History of chronic liver disease or suspected alcohol abuse
* Serum bilirubin greater than upper limit of normal unless attributable to Gilberts syndrome or haemolysis
* Alanine and/or aspartate aminotransferase levels (ALT and/or AST) and alkaline phosphatase (ALP) greater than 2.5 times the upper limit of normal
* Glomerular filtration rate (GFR) < 30ml/min. GFR calculated by Cockroft-Gault (not eGFR).
* Serological evidence of active hepatitis B or C infection whether acute or chronic (defined as positive anti-HCV serology; positive HBsAg). All positive HBcAb results should also be excluded on safety grounds regardless of HBsAg or HBV DNA status. Antibodies to Hepatitis B surface antigen (anti-HBs) due to a history of past vaccination is acceptable
* Known history of HIV seropositive status
* Patients with a history of Venoocclusive Disease (VOD) and Sinusoidal Obstructive Syndrome (SOS)
* Patients with a screening of QTcF interval >470msec
* Medical or psychiatric conditions compromising the patient's ability to give informed consent
* Women who are pregnant or lactating
* LVEF > 50% in the absence of significant co-morbidities that preclude anthracycline use
* Patients with a history of severe allergic/anaphylactic reaction to any humanised monoclonal antibody
* Patients with serious active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival | At 2 years following date of randomisation.
  Progression free survival rate and will be analysed using Kaplan-Meier survival analysis. PFS time will be measured from date of randomisation until progression or death.

SECONDARY OUTCOMES:
Overall response rate | Approximately 6 months after treatment start
  At the end of treatment
Overall Survival | 5 years from date of registration
  Date of registration until death.
Treatment toxicity | 7 months from beginning of treatment
  During treatment and follow up visits
Quality of life of patients during and after treatment | Baseline, during treatment and 6 month and 2 year follow up
  QoL questionnaires (EORTC QLQ-C30; Quality of life of cancer patients; 30 questions) to be completed by patient at time points listed below
Activities of Daily Living of patients during and after treatment | Baseline, during treatment and 6 month and 2 year follow up
  Activities of Daily Living questionnaire (ADL) to be completed by patient at time points listed below (6 questions about ability to undertake self-care)
Instrumental Activities of Daily Living of patients during and after treatment | Baseline, during treatment and 6 month and 2 year follow up
  Instrumental Activities of Daily Living questionnaire (IADL) to be completed by patient at time points listed below (8 questions about ability to undertake daily activities/self-care)
Performance status post treatment | Baseline, every 21 days for 8 cycles, 5 1/2 months at the end of treatment and then up to 3 years after the end of treatment.
  Performance status to be measured by investigator at time points listed below
Co-morbidities of patients | Baseline
  Details of co-morbidities to be recorded at point of randomisation by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McMillan, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (40):
- United Kingdom (40):
  - Stoke Mandeville Hospital (including Wycombe Hospital), Aylesbury
  - North Hampshire Hospital, Basingstoke
  - Royal United Hospital, Bath
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Oncology Centre, Bristol
  - West Suffolk Hospital, Bury St Edmunds
  - Kent and Canterbury Hospital, Canterbury
  - Castle Hill Hospital, Cottingham
  - University Hospital, Coventry, Coventry
  - Darent Valley Hospital, Dartford
  - Royal Devon & Exeter Hospital, Exeter
  - Medway Maritime Hospital, Gillingham
  - Beatson West of Scotland Cancer Centre (including Gartnavel Royal Hospital), Glasgow
  - James Paget University Hospital, Great Yarmouth
  - Northwick Park Hospital, Harrow
  - Kettering General Hospital, Kettering
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Aintree University Hospital, Liverpool
  - Royal Liverpool University Hospital, Liverpool
  - Guy's Hospital (including St Thomas's Hospital), London
  - Royal Free Hospital, London
  - University College London Hospital, London
  - Luton and Dunstable Hospital, Luton
  - Christie Hospital, Manchester
  - Freeman Hospital, Newcastle
  - North Tyneside Hosptial (including Wansbeck Hospital and Hexham General Hospital), North Shields
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Princess Royal University Hospital, Orpington
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Queen's Hospital, Romford
  - Southampton General Hospital, Southampton
  - Kings Mill Hospital, Sutton in Ashfield
  - Torbay Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - Royal Hampshire County Hospital, Winchester
  - Worcester Royal Hospital (including Kidderminster Hospital and Alexandra Hospital), Worcester
  - Wythenshawe Hospital (including Trafford General Hospital), Wythenshawe